CLINICAL TRIAL: NCT04189679
Title: : Identification of a Predictive Metabolic Signature of Response to Immune Checkpoint Inhibitors in Non-Small Cell Lung Carcinoma
Brief Title: Identification of a Predictive Metabolic Signature of Response to Immune Checkpoint Inhibitors in Non-Small Cell Lung Carcinoma
Acronym: METABO-ICI
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC19.133; 2019-A01255-52 (Other: ID RCB)
Record Dates: First submitted 2019-10-03; First posted 2019-12-06 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Metabolomic; Microbiota
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Meta-genomic signature of intestinal flora
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- First line: 20 patients in first line of treatment
  Interventions: Other: Immune signature in serum associated to the metabolic signature; Genetic: Meta-genomic signature of intestinal flora
- Second or third line: 40 patients in second and third line of treatment
  Interventions: Other: Immune signature in serum associated to the metabolic signature; Genetic: Meta-genomic signature of intestinal flora

INTERVENTIONS:
Other: Immune signature in serum associated to the metabolic signature — Immune signature in serum associated to the metabolic signature
Genetic: Meta-genomic signature of intestinal flora — Meta-genomic signature of intestinal flora

SUMMARY:
Immune checkpoints inhibitors (ICI) are becoming new standards of care for Non-Small Cell Lung Carcinoma (NSCLC) treatment. To date, no powerful predictive biomarker of response has been found.

The investigators hypothesize that metabolomics profile could represent a potent biomarker of response to ICI

DETAILED DESCRIPTION:
Immune checkpoints inhibitors (ICI) are becoming new standards of care for Non-Small Cell Lung Carcinoma (NSCLC) treatment, both as first and second line of treatment. To date, no powerful predictive biomarker of response has been found. It has been recently shown that microbiota composition could dictate the ability of patients to respond to ICI. Since, the microbiota produces circulating metabolites that will subsequently act on immune system, the investigators hypothesized that metabolic signature, reflecting microbiota function, could represent a predictive biomarker of response to ICI.

Primary objective is to identify baseline metabolic signature (metabolomics analysis by Mass spectrometry) associated to ICI response. Secondary objectives are to link metabolic signature with microbiota composition (metagenomics analysis RNA 16S) and immune profile, and altogether with clinic response to ICI. Profile evolution (metabolic, metagenomics and immune) will be also analyzed at 2-month post ICI initiation and at tumor progression, if any.

In order to do so, the investigators thus plan to enroll 60 NSCLC patients treated by ICI as 1st, 2nd or 3rd line of treatment in CHUGA in 18 months. Blood as well feces will be collected prior to, and at 2 month following ICI treatment initiation as well as at progression. Will be excluded from this study, patients that have received antibiotic or corticotherapy 2 or 4 weeks before ICI initiation, respectively.

ELIGIBILITY:
Inclusion Criteria:

* NSCLC diagnosis
* Patient treated by a ICI in first, second or third line of treatment, or by the combination of chemotherapy and IPCI in first line of treatment
* Patient with at least one measurable lesion as defined by RECIST

Exclusion Criteria:

* Patient treated with antibiotic treatment within 2 weeks before the start of ICI or corticosteroids (>20 mg per day) within 4 weeks before the start of ICI

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study cohort will include NSCLC patients treated by ICI as 1st, 2nd or 3rd line of treatment in Grenoble University Hospital (France) in 18 months. 60 NSCLC patients are anticipated to be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2020-01-03 (Actual); Primary Completion 2023-01-27 (Actual); Study Completion 2023-01-27 (Actual)

PRIMARY OUTCOMES:
Identification of the change from baseline Metabolic signature as predictive factor of the ICI response at 6 months or at the tumoral progression | baseline, 6 months or tumoral progression
  To identify the link of the change from baseline of Metabolic signature in serum (metabolomics analysis performed using a Mass spectrometry) and the ICI response at 6 months or at the tumoral progression

SECONDARY OUTCOMES:
Identification of the link between the Meta-genomic and immune signatures and the metabolic signature at 6 months or at the tumoral progression | 6 months or tumoral progression
  To identify the link between the Meta-genomic signature of intestinal flora (microbiota composition analysed by RNA 16 S) with the Immune signature in serum and the metabolic signature at 6 months or at the tumoral progression
Identification of the link between the Meta-genomic and immune signatures and ICI response at 6 months or at the tumoral progression | 6 months or tumoral progression
  To identify the link between the Meta-genomic signature of intestinal flora with the Immune signature in serum and the ICI response at 6 months or at the tumoral progression
Description of the profile change of Meta-genomic signature | 2 months or tumoral progression
  To describe the change from baseline of the Meta-genomic signature at 2 months or at the tumoral progression
Description of the profile change of Immune signature at 2 months or at the tumoral progression | Baseline and 2 months or tumoral progression
  To describe the change from baseline of the Immune signature at 2 months or at the tumoral progression
Identification of the link between the profile change of meta-genomic signature and the ICI response at 2 months or at the tumoral progression | Baseline and (2 months or tumoral progression)
  To identify the link between the profile change from baseline of meta-genomic signature and the ICI response at 2 months or at the tumoral progression
Identification of change of immune signature and the ICI response at 2 months or at the tumoral progression | Baseline and (2 months or tumoral progression)
  To identify the link between the profile change from baseline of immune signature and the ICI response at 2 months or at the tumoral progression
Description of overall survival under ICI at 6 months or at the tumoral progression | 6 months or tumoral progression
  To describe of the overall survival under ICI at 6 months or at the tumoral progression
Description of the survival without progression under ICI at 6 months or at the tumoral progression | 6 months or tumoral progression
  To describe the survival without progression under ICI at 6 months or at the tumoral progression

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Claire Toffart, Dr, Principal Investigator — University Hospital, Grenoble; Dalil Hannani, PhD, Study Director — Medicine University, Grenoble
Locations (1):
- University Hospital, Grenoble, La Tronche, Isère, France

IPD SHARING:
Plan to Share IPD: No